CLINICAL TRIAL: NCT07149233
Title: Effectiveness of Inspiratory Muscle Training on Objective and Subjective Sleep Parameters in Patients With Obstructive Sleep Apnea: A Randomized Controlled Trial
Brief Title: Effectiveness of Inspiratory Muscle Training on Sleep in Patients With Obstructive Sleep Apnea
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, shirley nogueira de souza, MSc student in Physical Therapy,Principal Investigator, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 7.330.179; CAAE: 84723724.2.0000.5208 (Other: Federal University of Pernambuco)
Record Dates: First submitted 2025-06-06; First posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Obstructive Sleep Apnea (OSA); Sleep
Keywords: Obstructive Sleep Apnea; Inspiratory Muscle Training; Objective and Subjective Sleep Parameters
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Intervention Model Description: Eligible participants will be assessed before and after four weeks of Inspiratory Muscle Training (IMT). Data will be recorded in evaluation forms covering personal, clinical, anthropometric variables, and respiratory muscle strength and performance. Participants will complete the Epworth Sleepiness Scale, Pittsburgh Sleep Quality Index, and International Physical Activity Questionnaire. Objective sleep data will be collected via actigraphy for nine days pre- and post-intervention, recorded in actigraphy forms. Nocturnal oximetry and polygraphy will also be performed before and after IMT, during the same weeks as actigraphy, and documented accordingly. IMT adherence will be self-reported in an IMT diary. After completing the intervention, participants will answer a questionnaire assessing perceived health changes and satisfaction with the treatment
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 - Inspiratory Muscle Training (IMT) (Experimental): Participants with moderate to severe obstructive sleep apnea (OSA) will perform inspiratory muscle training using a threshold device with progressive loading over 4 weeks. Training will begin at 50% of maximal inspiratory pressure (MIP) for the first 2 weeks, increase to 60% in week 3, and 75% in week 4. Participants will perform three sets of 30 fast, forceful inspiratory efforts, with one-minute rest intervals between sets. Training sessions will occur twice daily, seven days per week. Load adjustments will be made weekly during in-person visits. Participants will record adherence and occurrences in a training diary and will be monitored daily by the principal investigator through phone calls.
  Interventions: Device: Inspiratory Muscle Training
- Group 2 - Sham Inspiratory Muscle Training (Sham Comparator): Participants in the control group will perform sham inspiratory muscle training using the same device with the internal spring removed, providing no resistance. The training protocol will mirror that of the intervention group: three sets of 30 fast inspiratory efforts, with one-minute rest intervals, performed twice daily, seven days per week, for 4 weeks. Weekly in-person visits will be held to verify procedures, and participants will log adherence in a training diary. Daily phone follow-ups will be conducted by the principal investigator.
  Interventions: Device: Inspiratory Muscle Training

INTERVENTIONS:
Device: Inspiratory Muscle Training — Inspiratory muscle training (IMT) was performed for 4 weeks in patients with moderate to severe OSA. The intervention group used a threshold device with resistance: training occurred twice daily, 7 days per week, with 3 sets of 30 fast inspiratory efforts and 1-minute rest between sets. Load started at 50% of maximal inspiratory pressure (MIP), increased to 60% in week 3, and 75% in week 4. Weekly visits were held for load adjustment. The sham group followed the same schedule using the same device without resistance (spring removed). Both groups recorded adherence in training diaries and received daily follow-up calls from the principal investigator

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness of inspiratory Muscle Training (IMT) on both objective and subjective sleep parameters in patients with OSA.Methods: A prospective, randomized, controlled clinical trial will be conducted with patients diagnosed with OSA followed at Otavio de Freitas Hospital. Participants will be evaluated for excessive daytime sleepiness (Epworth Sleepiness Scale), sleep quality (Pittsburgh Sleep Quality Index), physical activity level (IPAQ), sleep latency, total sleep time, sleep efficiency, number of nocturnal awakenings, total time in bed, total wake time during sleep (Actigraphy), hypoxic burden during sleep (Nocturnal Oximetry), disease severity (Polysomnography), respiratory muscle strength (Manovacuometry), and respiratory muscle endurance (Powerbreathe K-series) before and after 4 weeks of training, as well as perceived change in health status after IMT (PGIC).Participants will be divided into two groups and will perform IMT for 4 weeks: the experimental group will perform IMT with a progressive weekly load (50%, 60%, 75% of MIP) adjusted using the Powerbreathe® Classic device, while the control group will use the device without load. The participants will perform IMT at home under the guidance of the principal investigator.Statistical Analysis: Data will be analyzed using SPSS version 26.0 with descriptive and analytical statistical techniques. Normality will be assessed using the Shapiro-Wilk test. For intergroup and intragroup comparisons, two-way ANOVA will be used. Tukey's post-hoc test will be applied to compare pre- and post-intervention mean variances for each group. The level of significance adopted for all analyses will be 95% (p < 0.05).Expected Results: It is expected that 4 weeks of IMT in patients with OSA will reduce excessive daytime sleepiness, sleep latency, number of awakenings, and hypoxic burden, as well as increase sleep efficiency and total sleep time, leading to improved sleep quality.

DETAILED DESCRIPTION:
Obstructive Sleep Apnea (OSA) is a prevalent sleep-related breathing disorder characterized by repeated episodes of upper airway obstruction during sleep, leading to intermittent hypoxia, sleep fragmentation, and frequent arousals. These events disrupt sleep architecture, reduce total sleep time and sleep efficiency, and result in non-restorative sleep. As a consequence, patients often present with excessive daytime sleepiness, cognitive and functional impairments, and an increased risk of occupational errors and motor vehicle accidents.

The impact of OSA extends beyond sleep, contributing to reduced quality of life and increased cardiovascular and metabolic risks. Considering the multifactorial consequences of OSA and the barriers to continuous positive airway pressure (CPAP) adherence-including cost, discomfort, and access-there is a need for alternative or adjunctive low-cost therapies that are easy to implement and have proven efficacy.

Inspiratory Muscle Training (IMT) has emerged as a promising therapeutic strategy to improve respiratory muscle strength, reduce symptoms, and potentially enhance sleep quality. However, evidence regarding its impact on objective and subjective sleep parameters in patients with OSA remains limited.

This study aims to evaluate the efficacy of a 4-week IMT protocol, following standardized training guidelines, in adults with moderate to severe OSA who have not yet initiated CPAP therapy. Validated instruments will be used to assess sleep outcomes. The findings are expected to contribute to clinical decision-making and offer evidence for non-pharmacological, non-invasive interventions to improve sleep quality and reduce daytime symptoms in this population.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants
* Age between 18 and 70 years
* Clinical diagnosis of moderate to severe Obstructive Sleep Apnea (OSA), confirmed by polysomnography
* Not currently undergoing treatment for OSA

Exclusion Criteria:

* Presence of neuromuscular disorders, infectious diseases, immunological conditions, tumors, or any disease that prevents inspiratory muscle training (IMT), manovacuometry, or respiratory muscle performance assessment
* Unstable angina, untreated or uncontrolled systemic arterial hypertension, left ventricular dysfunction, cerebral aneurysm, or any cardiovascular condition contraindicating IMT or respiratory muscle testing
* Upper limb deformities that prevent the use of actigraphy devices or oximetry sensors
* Other sleep disorders (e.g., insomnia, hypoventilation syndrome, or need for continuous home oxygen therapy)
* Cognitive impairment that limits the participant's ability to understand or follow study procedures
* Ongoing or planned CPAP therapy during the follow-up period
* Participation in a pulmonary rehabilitation program within 6 months prior to the study
* Moderate or high physical activity level according to the IPAQ, including regular moderate or vigorous physical activity within the past 30 days
* Use of sleep-inducing medication to treat insomnia
* Grade 2 or 3 obesity (BMI ≥ 35 kg/m²)
* Residence in a geographic area with limited or no access to telephone or internet service, preventing contact or data transmission from study devices (actigraphy and/or oximetry sensors)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-03-11 (Actual); Primary Completion 2025-12-20 (Estimated); Study Completion 2026-02-20 (Estimated)

PRIMARY OUTCOMES:
sleep quality | Sleep quality will be assessed before and after four weeks of inspiratory muscle training
  Sleep quality will be assessed using the PSQI. A score from 0 to 4 indicates good sleep quality, while a score above 5 indicates poor sleep quality
daytime sleepiness | Daytime sleepiness will be assessed before and after four weeks of inspiratory muscle training
  Daytime sleepiness will be assessed using the Epworth Sleepiness Scale (ESS) before and after the four weeks of inspiratory muscle training (IMT). The scale consists of eight everyday situations, asking the individual to self-assess the likelihood of dozing off during these activities, scoring from 0 to 3, where 0: no chance of dozing, 1: slight chance, 2: moderate chance, and 3: high chance. A total score greater than 10 is used as the cutoff point to identify individuals with a high likelihood of excessive daytime sleepiness

SECONDARY OUTCOMES:
hypoxic burden | The hypoxic burden will be assessed before and after four weeks of inspiratory muscle training
  To assess peripheral oxygen saturation (SpO2) levels during sleep, a sleep study will be conducted using a high-resolution wireless pulse oximeter. The collected data are automatically transferred to a cloud service where they are analyzed by an algorithm.
Maximal Inspiratory Pressure (MIP) | Baseline, weekly during intervention (for load adjustment), and post-intervention (4 weeks)
  Inspiratory muscle strength assessed by POWERbreathe KH2 in testing mode. The evaluation will be performed weekly during the intervention period to adjust training loads, and at baseline and post-intervention for analysis purposes; Unit of measure: cmH₂O
  ; Assessment tool: POWERbreathe KH2/K5
Disease severity | Disease severity will be assessed before and after four weeks of inspiratory muscle training.
  Disease severity will be assessed through polygraphy before and after the four weeks of inspiratory muscle training (IMT) in the study participants. The ApneaLink device (ResMed) will be used to evaluate disease severity
Physical activity level | Assessment Before and after 4 weeks
  Physical activity level will be assessed using the International Physical Activity Questionnaire (IPAQ), an instrument that estimates weekly energy expenditure from physical activities related to work, transportation, household tasks, and leisure.The IPAQ classification divides and defines physical activity levels into the following categories: low, moderate, or high
Respiratory endurance | Assessment Before and after 4 weeks
  Unit of measurement: (cmH₂O); Assessment tool: Powerbreathe KH2/K5
Fatigue Index Strength | Assessment Before and after 4 weeks
  Unit of measurement: (cmH₂O); Assessment tool: Powerbreathe KH2/K5
Peak inspiratory flow | Assessment Before and after 4 weeks
  Unit of measurement: (liters/second); Assessment tool: Powerbreathe KH2/K5
Energy inspiratory | Assessment Before and after 4 weeks
  Unit of measurement: (joules); Assessment tool: Powerbreathe KH2/K5
Volume inspiratory | Assessment Before and after 4 weeks
  Unit of measurement: (liters); Assessment tool: Powerbreathe KH2/K5
Bedtime | 9 days before the start of IMT and 9 days after completion of the 4-week IMT protocol
  Bedtime assessed objectively by actigraphy; Unit of measure: hours ;Assessment tool: ActTrust actigraph (Condor Instruments, Brazil)
Wake-up time | 9 days before the start of IMT and 9 days after completion of the 4-week IMT protocol
  Wake-up time assessed objectively by actigraphy; Unit of measure: hours; Assessment tool: ActTrust actigraph (Condor Instruments, Brazil)
Sleep latency | 9 days before the start of IMT and 9 days after completion of the 4-week IMT protocol
  nterval between bedtime and sleep onset measured by actigraphy.
  nterval between bedtime and sleep onset measured by actigraphy; Unit of measure: minutes (min); Assessment tool: ActTrust actigraph (Condor Instruments, Brazil)
Sleep efficiency | 9 days before the start of IMT and 9 days after completion of the 4-week IMT protocol
  Percentage of total sleep time (TST) divided by time in bed (TIB), derived from actigraphy; Unit of measure: percentage (%); Assessment tool: ActTrust actigraph (Condor Instruments, Brazil)
Total sleep time (TST) | 9 days before the start of IMT and 9 days after completion of the 4-week IMT protocol
  Total time spent asleep measured by actigraphy; Unit of measure: hours (h); Assessment tool: ActTrust actigraph (Condor Instruments, Brazil)
Time in bed (TIB) | 9 days before the start of IMT and 9 days after completion of the 4-week IMT protocol
  Total time in bed measured by actigraphy; Unit of measure: hours (h);
  Assessment tool: ActTrust actigraph (Condor Instruments, Brazil)
Number of awakenings after sleep onset | 9 days before the start of IMT and 9 days after completion of the 4-week IMT protocol
  Number of awakenings after sleep onset measured by actigraphy; Unit of measure: count (n); Assessment tool: ActTrust actigraph (Condor Instruments, Brazil)
Number of secondary sleep episodes after sleep onse | 9 days before the start of IMT and 9 days after completion of the 4-week IMT protocol
  Number of additional sleep episodes after initial sleep onset measured by actigraphy; Unit of measure: count (n); ssessment tool: ActTrust actigraph (Condor Instruments, Brazil)
Wake after sleep onset (WASO) | 9 days before the start of IMT and 9 days after completion of the 4-week IMT protocol
  Minutes of wakefulness after sleep onset measured by actigraphy; Unit of measure: minutes (min); Assessment tool: ActTrust actigraph (Condor Instruments, Brazil)
Maximal Expiratory Pressure (MEP) | Assessment Before and after 4 weeks
  Maximum expiratory pressure at the mouth during a maximal effort against occluded airway; Unit of measure: cmH₂O
  Assessment tool: HOMED MVD300 digital manovacuometer

CONTACTS AND LOCATIONS:
Overall Officials: Armele D de Andrade, PhD Pneumo, Study Director — Universidade Federal de Pernambuco
Locations (1):
- Cardiopulmonary Physiotherapy Laboratory, Recife, Pernambuco, Brazil

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) will be shared upon reasonable request for academic and research purposes, following approval by the principal investigator and compliance with ethical standards. Participants' privacy and confidentiality will be strictly maintained
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will be available beginning 6 months after publication of the primary study results, for a period of up to 5 years.
Access Criteria: Researchers must submit a detailed research proposal and obtain approval from the principal investigator.
URL: https://plataformabrasil.saude.gov.br

REFERENCES:
- [Background] Aiello KD, Caughey WG, Nelluri B, Sharma A, Mookadam F, Mookadam M. Effect of exercise training on sleep apnea: A systematic review and meta-analysis. Respir Med. 2016 Jul;116:85-92. doi: 10.1016/j.rmed.2016.05.015. Epub 2016 May 21. PMID 27296826
- See also: Brazilian platform for research project submission — https://plataformabrasil.saude.gov.br

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-12-30): https://cdn.clinicaltrials.gov/large-docs/33/NCT07149233/Prot_SAP_ICF_000.pdf